CLINICAL TRIAL: NCT06905639
Title: Impact of Physical Exercise on Lymphedema Related to Breast Cancer: Assessment Using Thermography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Arias Crespo (Other)
Collaborators: University of Leon (Unknown)
Responsible Party: Sponsor-Investigator, Marta Arias Crespo, Graduate in nursing, Universidad de León
Organization: Universidad de León (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETICA-ULE-055-2024; No aplicable (Other: No tiene)
Record Dates: First submitted 2025-03-12; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasms; Lymphedema; Thermography; Exercise
Keywords: Breast Neoplasms; Lymphedema; Exercise; Thermography
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a parallel-design interventional clinical study, in which participants will be randomly assigned to two groups. The first group will receive the intervention, which consists of a supervised physical exercise program, while the second group (control group) will continue with their usual routine of daily activities without additional intervention. Both groups will be evaluated throughout the study to compare the effects of physical exercise on the improvement or prevention of post-breast cancer lymphedema
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION GROUP (Experimental): This arm of the study consists of participants who will receive a supervised physical exercise intervention specifically designed to improve post-breast cancer lymphedema. The program includes a combination of strength exercises and aerobic exercises, aimed at improving mobility, reducing injury, and increasing muscle strength in the arm affected by lymphedema
  Interventions: Behavioral: Aerobic and Strength Exercise
- CONTROL GROUP (No Intervention): This arm of the study includes participants who will not receive any exercise intervention. They will continue with their usual daily routine and will be monitored throughout the study to compare changes in lymphedema between the intervention group and the control group

INTERVENTIONS:
Behavioral: Aerobic and Strength Exercise — A supervised physical exercise intervention was carried out, specifically designed to improve post-breast cancer lymphedema. The program will include a combination of strength exercises and aerobic exercises, with the aim of improving mobility, reducing inflammation, and increasing muscle strength in the arm affected by lymphedema
  Arms: INTERVENTION GROUP

SUMMARY:
Study Type: Clinical Trial

Primary Purpose: To determine whether physical exercise improves or prevents lymphedema in breast cancer patients.

Description of the Participant Population/Main Condition: The study is aimed at women who have been diagnosed with breast cancer and have experienced post-treatment lymphedema or are at risk of developing it. The target population includes adults aged 18 to 70 who have been diagnosed with this condition following their breast cancer treatment.

Main Research Questions:

Does physical exercise improve or prevent lymphedema in women with breast cancer? What are the effects of physical exercise on the reduction of arm volume affected by lymphedema? What are the effects of physical exercise on the reduction of perceived disability in the arm affected by lymphedema?

Hypothesis:

Physical exercise intervention significantly reduces lymphedema symptoms, such as arm volume. Physical exercise prevents the progression of lymphedema in women with breast cancer.

Comparison Group: Researchers will compare results between the experimental group (which will undergo physical exercise) and the control group (which will receive no intervention) to determine if physical exercise has a significant impact on the improvement or prevention of lymphedema.

Participant Tasks:

The experimental group will follow a supervised physical exercise program for a specific period. The control group will receive no intervention and will be monitored with standard follow-up care without exercise. Participants will be evaluated before and after the study period to measure the progression of lymphedema, including arm volume measurement and surface skin temperature using thermography.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old diagnosed with breast cancer.
* Residing in the province of León.
* Not currently undergoing any physical exercise intervention at the time of the study.
* Not participating in lifestyle modification programs at the time of the study.
* Not presenting any relative or absolute sequelae from chemotherapy treatment that would pose a relative or absolute contraindication to their participation in this intervention (e.g., cardiological sequelae).
* Having signed the informed consent to participate in the study.

Exclusion Criteria:

* Presenting physical and/or psychological limitations that would hinder understanding or the ability to carry out the established intervention program.
* Presenting an infection in the upper limbs or lymphangitis.
* Fluid accumulation in the breast area requiring drainage at the time of the intervention.
* Not having signed the informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Perimeters | 10 weeks
  The perimeter of the arm affected by lymphedema will be measured to assess the reduction in lymphedema volume in the participants. This measurement will be taken before and after the intervention to compare changes and determine the impact of physical exercise on inflammation and the size of the affected arm
Thermography | 10 weeks
  Thermography will be used to assess the temperature distribution in the arm affected by lymphedema. A thermal image will be taken before and after the intervention to observe changes in inflammation and circulation in the affected area, allowing the evaluation of whether physical exercise has an effect on the reduction of temperature associated with lymphedema
Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | 10 weeks
  The Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire will be used to assess the functionality of the arm in the participants. This questionnaire measures limitations in daily activities related to the arm affected by lymphedema. It will be administered before and after the intervention to assess changes in mobility and functional capacity following physical exercise. In the DASH questionnaire, higher scores indicate greater disability, while lower scores indicate less disability

SECONDARY OUTCOMES:
Bicipital and Tricipital Skinfolds | 10 weeks
  Bicipital and tricipital skinfold measurements will be taken to assess the body composition and body fat percentage of the participants. These measurements will help analyze the impact of physical exercise on the reduction of body fat and potential improvements in muscle mass, especially in the area affected by lymphedema. The skinfolds will be measured in millimeters (mm), and body fat percentage will be measured in percentage (%).
RS-14 Questionnaire (Resilience Scale for Adults) | 10 weeks
  The RS-14 Questionnaire (Resilience Scale for Adults) will be used to assess resilience in the participants. This questionnaire will allow us to observe whether the physical exercise intervention has an effect on the participants. In the RS-14 questionnaire, higher scores indicate greater resilience, while lower scores indicate lower resilience.
  Maximum and Minimum Scores: The questionnaire consists of 14 items, each rated on a Likert scale from 1 to 7, where:
  1 means "strongly disagree" 7 means "strongly agree"
  The scores are summed to obtain a total score, with a scoring range of 14 to 98:
  Minimum score: 14 (low resilience) Maximum score: 98 (high resilience)
Trait Meta-Mood Scale (TMMS-24) | 10 weeks
  The Trait Meta-Mood Scale (TMMS-24) questionnaire will measure the level of emotional intelligence in the participants, including the perception, understanding, and regulation of emotions. It will be administered before and after the intervention to evaluate whether physical exercise influences the improvement of emotional intelligence in patients with lymphedema.
  Scores: The TMMS-24 questionnaire consists of 24 items, distributed across three dimensions:
  Emotional Perception Emotional Understanding Emotional Regulation
  Each item is rated on a Likert scale from 1 to 5, where:
  1 means "strongly disagree" 5 means "strongly agree"
  Scores are summed within each dimension, and a total emotional intelligence score is obtained, with score ranges indicating different levels of emotional ability:
  Low score: Indicates lower capacity in emotional perception, understanding, and regulation.
  High score: Indicates greater capacity in these areas.
MOS Social Support Survey (MOS-SSS) | 10 weeks
  The MOS Social Support Survey (MOS-SSS) questionnaire will be used to measure the level of social support received by the participants. This questionnaire will help identify how social support may influence the response to physical exercise.
  Scores: The MOS-SSS questionnaire consists of several questions related to different dimensions of social support, such as emotional, instrumental, and relational support. Responses are rated on a Likert scale from 1 to 5, where:
  1 means "None" (indicating a very low level of social support) 5 means "A lot" (indicating a very high level of social support) Scores are summed to obtain a total score, and in this case, higher scores indicate a higher level of social support, while lower scores indicate a lower level of social support.
Anthropometric measurements | 10 weeks
  Changes in the participants' weight will be evaluated throughout the study. Weight will be measured in kilograms (kg), and these measurements will allow us to observe whether the physical exercise intervention has an effect on weight loss or gain in the participants. Additionally, the Body Mass Index (BMI) will be calculated for each participant, which is obtained by dividing weight (in kilograms) by height squared (in meters). The height of the participants will also be measured in meters (m) to assess changes in their overall body composition.
Percentage of water | 10 weeks
  Body water percentages will be measured for each participant using validated measuring devices, such as a Tanita. This will provide a more complete picture of changes in body composition, as body water is a key indicator of hydration and overall body balance. With these measurements, it will be possible to identify variations in the distribution of fluids and other important components of the body over time.
Percentage of fat | 10 weeks
  Body fat percentages will be measured for each participant using validated measuring devices, such as a Tanita. This will provide a more complete picture of changes in body composition, as body water is a key indicator of hydration and overall body balance. With these measurements, it will be possible to identify variations in the distribution of fluids and other important components of the body over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de León, Ponferrada, León, Spain

IPD SHARING:
Plan to Share IPD: No